CLINICAL TRIAL: NCT04726098
Title: Efficacy of Low or High Dose of Dexamethasone in Patients With Respiratory Failure by COVID-19
Brief Title: Low or High Dose of Dexamethasone in Patients With Respiratory Failure by COVID-19
Acronym: HIGHLOWDEXA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Manuel Taboada Muñiz (Other)
Responsible Party: Sponsor-Investigator, Manuel Taboada Muñiz, Associate Proffesor, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIGHLOWDEXA-COVID; 2020-005702-25 (EudraCT Number)
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Corticosteroids
Keywords: COVID19; respiratory failure; corticosteroids
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label trial involving hospitalized adult patients with respiratory failure needing oxygen therapy, caused by COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose group (Active Comparator): Dexamethasone 6mg/day for 10 days
  Interventions: Drug: Dexamethasone low dose
- High dose group (Active Comparator): Dexamethasone 20mg/day for 5 days + Dexamethasone 10mg/day for 5 days (Total 10 days)
  Interventions: Drug: Dexamethasone high dose

INTERVENTIONS:
Drug: Dexamethasone high dose — High doses: dexamethasone 20 mg/day 5 days + 10 mg/day 5 days (total 10 days)
  Arms: High dose group
Drug: Dexamethasone low dose — Low doses: dexamethasone 6 mg/day 10 days.
  Arms: Low dose group

SUMMARY:
After RECOVERY trial publication, low dose (6 mg dexamethasone for 10 days) was recommended as the usual care treatment in hospitalized patients with respiratory failure by COVID-19 needing oxygen therapy. RECOVERY trial showed how the use of dexamethasone 6 mg / day for ten days compared to standard treatment without the use of corticosteroids in hospitalized patients reduced mortality at 28 days (22.9% with dexamethasone vs 25.7% without dexamethasone). In the dexamethasone group, the incidence of mortality was lower than standard treatment in patients with hypoxia and the need for mechanical ventilation (29.3% with dexamethasone vs 41.4% without dexamethasone), in patients admitted to the hospital ward with a need for oxygen therapy (23.3% with dexamethasone vs 26.2% without dexamethasone), but they did not find differences between those admitted patients who did not need oxygen therapy. There are two other studies (DEXA-COVID-19 and CoDEX) where they observed benefits of the use of dexamethasone 20 mg / day 5 days, and 10 mg / day 5 days (total 10 days) in patients admitted for respiratory distress syndrome (ARDS) and COVID-19. At present, it is unclear what dose of dexamethasone is most beneficial in patients with COVID-19 and respiratory failure.

DETAILED DESCRIPTION:
Objective: The investigators aim to assess the efficacy of high dose of dexamethasone (20 mg / day 5 days, and 10 mg/day 5 days) versus low dose of dexamethasone (6 mg/day 10 days) in patients with respiratory failure by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Hospitalized COVID-19 patients admitted to the Hospital.
* Patients requiring supplemental oxygen. Level 4 using the World Health Organization 7-point Ordinal Scale for clinical improvement
* Patients requiring corticosteroids (dexamethasone) according to Hospital protocol.

Exclusion Criteria:

* Pregnancy or active lactation.
* Patient is expected to die in the next 48 hours.
* Known history of dexamethasone allergy or known contraindication to the use of corticosteroids.
* Daily use of corticosteroids in the past 15 days.
* Indication for corticosteroids use for other clinical conditions (e.g. refractory septic shock).
* Consent refusal for participating in the trial.
* Different level of 4 in Level 4 using the World Health Organization 7-point Ordinal Scale for clinical improvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with treatment failure at day 11 | Day 11 after randomization
  defined as death, need of ICU and extracorporeal membrane oxygenation, need of non-invasive ventilation or nasal high-flow oxygen therapy, or worsening of the condition clinic of the patient during treatment (two of these: need to increase Fraction of inspired oxygen inspired>20%, need for fraction inspired oxygenation>50%, increase in respiratory rate>25, increase in inflammatory markers).

SECONDARY OUTCOMES:
Percentage of patients without the need for oxygen support at day 11. | Day 11 after randomization
28-days mortality | 28 days after randomization
90-days mortality | 90 days after randomization
Clinical status of patients using the World Health Organization 7-point Ordinal Scale for clinical improvement during 10 days of treatment | 10 days after randomization
  1:Not hospitalized, 2:Hospitalized and not treatment, 3: Hospitalized with treatment, not requiring supplemental oxygen, 4:Hospitalized requiring supplemental oxygen, 5:Hospitalized, requiring non-invasive ventilation or nasal high-flow oxygen therapy, 6: Hospitalized requiring invasive ventilation or Extracorporeal (ECMO)
Percentage of patients needing Intensive Care Unit admission | 28 days after randomization
Percentage of patients needing invasive mechanical ventilation or extracorporeal membrane oxygenation | 28 days after randomization
Percentage of patients needing non-invasive ventilation or nasal high-flow oxygen therapy | 28 days after randomization
Length of stay in the hospital | 90 days after randomization
Infectious complications during hospital admission | 90 days after randomization
Adverse drug reactions | 11 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada Muñiz, Ph.D., Principal Investigator — University Clinical Hospital of Santiago de Compostela
Locations (1):
- University Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taboada M, Rodriguez N, Varela PM, Rodriguez MT, Abelleira R, Gonzalez A, Casal A, Diaz Peromingo JA, Lama A, Dominguez MJ, Rabade C, Paez EM, Riveiro V, Pernas H, Beceiro MDC, Caruezo V, Naveira A, Carinena A, Cabaleiro T, Estany-Gestal A, Zarra I, Pose A, Valdes L, Alvarez-Escudero J. Effect of high versus low dose of dexamethasone on clinical worsening in patients hospitalised with moderate or severe COVID-19 pneumonia: an open-label, randomised clinical trial. Eur Respir J. 2022 Aug 4;60(2):2102518. doi: 10.1183/13993003.02518-2021. Print 2022 Aug. PMID 34916266